CLINICAL TRIAL: NCT05622773
Title: Anti-Fatigue Mat For Operating Room Nurses Fatigue And Bottom Of Use And Foot Bath Effect on Extremity Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neşe Uğur (Other)
Collaborators: Bartin State Hospital (Other Government); Bulent Ecevit University (Other)
Responsible Party: Sponsor-Investigator, Neşe Uğur, master degree student, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-SBB-0330
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Lower Extremity Pain; Fatigue
Keywords: operating room nurse; anti-fatigue mat; lower extremity; foot bath; fatigue; pain
MeSH Terms: conditions — Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: Pretest posttest single group quasi-experimental research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one-group quasi-experimental study (Experimental): Materials for Introductory Information Form, Visual Analog Scale (VAS), Visual Similarity Scale for Fatigue (VAS-F), Lower Leg Circumference Measurement Monitoring Form, Lower Extremity Edema Monitoring Form, Anti-Fatigue Mat, Foot Bath will be used in data collection. During the data collection process, the basic measurements of the operating room nurses will be made and then the measurements will be repeated using an anti-fatigue mat. The collection of data will be interrupted for 1 month, and basic measurements will be taken again and the nurses will be provided with a foot bath. After the footbath applications, the measurements will be repeated and recorded.
  Interventions: Other: Mat use application

INTERVENTIONS:
Other: Mat use application — In the research, repeated measurements will be made by using mats and foot baths in a single group and the data will be recorded.
  Other Names: Foot bath application

SUMMARY:
Summary Introduction: Prolonged standing brings with it various health problems such as extremity pain, fatigue, cardiovascular abnormalities. According to the Ergonomic Tool 4 guideline of the Perioperative Registered Nurses Association (AORN); If a staff member has to stand for more than two hours, stand in the same position for more than 30% of the working day or while wearing a lead apron, ergonomic intervention and alternative methods are recommended.

Purpose: The aim of this thesis study is to examine the effects of anti-fatigue mat use and footbath on fatigue and lower extremity pain among operating room nurses.

Method: This study, which was designed as a pretest posttest single-group quasi-experimental type, will be carried out with 27 nurses working in the operating room department between September 2022 and June 2023 at Bartın State Hospital, Bartın Gynecology and Childhood Diseases Hospital and Zonguldak Bülent Ecevit University Health Practice and Research Center. Introductory Information Form, Visual Analog Scale (VAS), Visual Similarity Scale for Fatigue (VAS-F), Lower Leg Circumference Monitoring Form, Lower Extremity Edema Monitoring Form, Anti-Fatigue Mat, Materials for Foot Bath will be used in data collection. During the data collection process, the basic measurements of the operating room nurses will be made and then the measurements will be repeated using an anti-fatigue mat. The collection of data will be interrupted for 1 month, and basic measurements will be taken again and the nurses will be provided with a foot bath. After the footbath applications, the measurements will be repeated and recorded. Data will be saved in SPSS 22.0 Program. In the evaluation of the data obtained, tests evaluating the normal distribution of the data will be used as well as descriptive statistical methods. According to the normal distribution of the data, the data will be analyzed with parametric or nonparametric tests.

Conclusion: At the end of the study, it is expected that there will be significant differences between the two applications in terms of fatigue, pain in the lower extremities and edema, and it will be beneficial. There are very few studies on the use of mats and foot baths in operating room nurses. There is no study evaluating the combined effect of both. It will be an example for the literature and future studies.

DETAILED DESCRIPTION:
Musculoskeletal disorders; It is defined as dysfunctions affecting various parts of the body, including muscles, bones, joints and spinal discs. These dysfunctions are mainly caused by repetitive manual work, lifting heavy loads, standing for long periods and working in fixed or inappropriate postures. Studies have shown that healthcare professionals (especially those working in operating rooms and intensive care units) face various problems related to long-term standing.

A person's body is affected by the conditions of his work area and his actions while standing. Keeping the body in an upright position requires significant muscle effort. Prolonged standing is one of the most common situations that requires muscle effort and causes various health problems. Prolonged standing significantly reduces blood flow to the muscles, accelerating the onset of fatigue in the extremities. It causes pooling of blood in the legs and feet, and pain in the lower extremities, back and neck muscles. When evaluated in terms of cardiovascular system; Carotid arteriosclerosis, leg edema, orthostatic symptoms (dizziness, etc.), changes in heart rate, blood pressure, and venous diseases (chronic venous insufficiency, etc.) can be observed in individuals. In addition, prolonged standing can cause temporary immobility of the joints in the spine, hips, knees and feet. This inactivity can then lead to rheumatic diseases due to degenerative damage to tendons and ligaments. Studies consistently report that the reporting of musculoskeletal disorders due to constant standing, such as low back pain, physical fatigue, myalgia, leg edema, fatigue, is increasing.

It is reported that musculoskeletal disorders cause labor losses and re-employment costs, especially in healthcare personnel, between 27,000-103,000 USD per nurse. The National Health System, the largest employer in the UK; It has a high rate of absenteeism from work due to illness due to musculoskeletal conditions, equivalent to around £400 million and 9.5 million working days per year. According to the German Federal Institute for Occupational Safety and Health, musculoskeletal disorders cause the highest cost compared to all other disease diagnostic groups. It causes a production loss of 17.2 billion euros and a gross value added loss of 30.4 billion euros per year. 5.43 million euro of these losses and 6.69 million euro of gross value added loss cover the public sector, including the education and health sector. Studies in Europe have shown that approximately 40 million workers are adversely affected by these ailments, accounting for 0.5-2% of the Gross Domestic Product of the European Union. Although musculoskeletal disorders have a high prevalence among communities around the world, healthcare professionals are faced with these problems more. The prevalence of musculoskeletal disorders has been reported to range from 40% to 90% among nurses worldwide. The prevalence of discomfort in the knees; It has been reported in five studies conducted in Iran, the USA, Switzerland and the Netherlands. According to the results of the random effects model, the prevalence of this disorder was determined as 43.43% (CI 95%: 23.80-63.06). In the ankles and feet, the prevalence was shown to be 57.06%. Study results reveal a high prevalence of musculoskeletal disorders among operating room personnel, especially in the lower back, back, neck, shoulders, ankles, and feet.In a study conducted at Cairo University on 184 operating room nurses, the most affected body parts of nurses in the last 12 years were the waist (76.1%), knees (67.9%), ankles/feet (60.9%) and neck (57.1%).In a study conducted in our country, it was found that 56.8% of musculoskeletal pain was in the back, 51.9% in the low back and 49.4% in the neck region in 162 operating room nurses; it was determined that these were followed by the shoulder (43.2%), foot/ ankle (38.3%) and knee (31.5%) regions, respectively.

According to AORN, operating room nurses encounter a variety of ergonomic stressors in their daily work. Job requirements for OR nurses may include lifting 25 kg on their own or 75 kg with assistance, the ability to work in an environment with unpleasant sights and smells, stressful situations, radiation, infection and hazardous materials. The AORN Workplace Safety Task Force began work in 2005 to identify high-risk ergonomic tasks. One of them is standing for long periods of time. Many OR nurses have to stand for long periods of time, which brings with it the risk of various health problems (eg extremity pain, cardiovascular abnormalities). AORN's Ergonomic Tool 4; ergonomic intervention is required if a staff member has to stand for more than two hours, stand in the same position for more than 30% of the workday, or while wearing a lead apron. In a study conducted in the United Kingdom to investigate the prevalence of pain experienced by 130 surgeons from various subspecialties of surgery, it was reported that the most common pain experienced by surgeons was low back pain, which in approximately 43% was severe enough to force interruption of surgery to relieve symptoms. In the study, foot pain also stands out as the type of pain that surgeons experience during surgery, but it is reported that surgeons have difficulty in finding suitable shoe recommendations.

While many surgeries that could not be performed due to COVID-19 are slowly returning, it is emerging that surgeons and operating room nurses need equipment and practices that support better ergonomics. Since the operating room is one of the most sensitive and valuable parts of hospitals, the operating room personnel should be given due care and appropriate ergonomic conditions should be provided. If measures are not taken to eliminate the discomfort, not only will employee health be adversely affected, but also the workflow in the operating room will be negatively affected. The AORN "Guideline for Safe Patient Transport and Movement 8" recommends the use of anti-fatigue mats in the operating room environment to counter the effects of prolonged standing. Anti-fatigue mat to reduce fatigue caused by prolonged standing on a hard surface. They are ergonomic structures designed for flexible surface. Fatigue-reducing mats can be made from various materials such as rubber, carpet materials, vinyl and wood. Anti-fatigue mats are often used to reduce lower extremity discomforts for workers who stay in the same position for long periods of time. They absorb static shock and reduce foot fatigue. However, it requires caution in the use of mats, as it may cause accidents such as tripping and falling. The use of non-slip mats should be preferred. It provides venous flow by stimulating muscle activation. It is beneficial in increasing foot comfort and safety.Operating room nurses stay up for one to eight hours during most of their shifts. To reduce the effects of the same position and standing for a long time; use of anti-fatigue mats, sit-stand stools, compression stockings, etc. It is recommended to use options. One study subjectively assessed low back pain in a standing position with a normal surface and on an anti-fatigue mat. The findings revealed that the anti-fatigue mat significantly reduced the subjective pain level in the lumbar region among the 15 participants (p < 0.05). However, it was concluded that the anti-fatigue mat does not objectively significantly alter the gluteus medius muscle activation associated with low back pain. In another study conducted on 127 surgeons; It has been determined that the use of mats reduces the feeling of discomfort in surgeons who experience fatigue, discomfort, stiffness and pain, but there is no significant difference in leg circumference change due to mat use.

In addition to ergonomic conditions, foot bath is one of the economical methods that has a positive effect on pain and fatigue in the lower extremities. Foot bath treatment is a complementary and alternative therapy that is effective in reducing fatigue and stress by stimulating the feet with warm water, accelerating blood circulation and metabolism from the capillaries under the skin, and stimulating the parasympathetic nerves. Foot bathing also has benefits such as reducing heart rate, improving sleep quality and body movement. In one study, keeping the feet of patients in warm water at 38-42 C for 20 minutes was found to be an effective approach to relieve pain. In a study conducted on nursing students in Korea, there was no evidence that footbathing was effective on fatigue levels, but it was determined that footbathing for two weeks had a positive effect on reducing leg edema. In the study on the subject, in the operating room nurses; Foot bathing has been found to reduce leg edema, physical stress and fatigue.

When the studies are examined, it is noteworthy that the studies evaluating the effectiveness of foot bath and anti-fatigue mat use in operating room nursing on fatigue and lower extremity disorders are limited.

ELIGIBILITY:
Inclusion Criteria:

* Working as a sterile nurse in the operating room
* Volunteering
* Don't be a smart phone
* No hearing or vision problems
* No diagnosed health problem in the lower extremities
* Working as a sterile nurse in the operating room for at least 4 hours a day
* Not using compression stockings

Exclusion Criteria:

* Working as a circulating nurse in the operating room
* Not willing to participate in research
* Have a diagnosed lower extremity problem
* Not having a smart phone
* Hearing and vision problems
* Using compression stockings

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Follow-up | It consists of a 4-week follow-up follow-up. Pain intensity will be evaluated separately for both feet before and after both applications.
  Visual Analog Skala (VAS)
Fatigue Follow-up | It consists of a 4-week follow-up follow-up. Fatigue severity will be evaluated before and after both applications.
  Visual Similarity Scale for Fatigue (VAS-F)
Lower Leg Circumference Measurement Follow-up | In the 4-week tables created, right and left calf; First, the measurements will be recorded before and after using the anti-fatigue mat for a month, and then before and after the footbath application.
  Lower Leg Circumference Measurement
Edema Follow-up | For edema monitoring, pressure is applied to the pretibial area for 5 seconds. The rating is from +1 to +4. ( 1 +): Slight gode is formed with pressure. (2mm) Gode returns in 15 seconds. (2++): Deep godet is formed with pressure. (4mm). Gode returns in
  Edema
mat use application | It will be collected just before the first shift of the week for a period of one month and 10 minutes after the end of the case after the use of the mat in the third shift.
  anti fatigue mat
Foot bath application | At 38-40 °C, it will be desirable to immerse both feet in water up to the ankle line for 20 minutes per day. All measurements will be collected and recorded just before the start of the first shift, 10 minutes after the end of the surgery and footbath in
  Foot bath

CONTACTS AND LOCATIONS:
Overall Officials: Sevim ÇELİK, Prof, Study Director — Bartin University Health Science Faculty; Neşe Uğur, Study Chair — Bartın Satate Hospital
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No